CLINICAL TRIAL: NCT01884298
Title: Effect of Different Anesthetic Techniques for Isolated Systolic Hypertensive Patients of Abdominal Surgery on Postoperative Hospital Stay and morbidity---a Prospective, Randomized Study
Brief Title: Effect of Different Anesthetic Techniques for Isolated Systolic Hypertensive Patients of Abdominal Surgery on Postoperative Hospital Stay and Morbidity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, ZhouYan, MD, Peking University First Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: EPIISO-021
Record Dates: First submitted 2013-06-19; First posted 2013-06-24 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Postoperative Complications
Keywords: remifentanil; isolated systolic hypertension; morbidity; epidural combined general anesthesia
MeSH Terms: conditions — Postoperative Complications; Isolated Systolic Hypertension | interventions — Remifentanil; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- patients with isolated systolic hypertension (Experimental): patients combined with isolated systolic hypertension undergoing abdominal surgery
  Interventions: Drug: remifentanil(Ultiva); Drug: epidural infusing 2% lidocaine

INTERVENTIONS:
Drug: remifentanil(Ultiva) — remifentanil (TCI, Ce 3 ng /ml)for intra-operative analgesia
Drug: epidural infusing 2% lidocaine — epidural infusing 2% lidocaine 4ml bolus followed by 6-18ml/hr for intra-operative analgesia

SUMMARY:
In General anesthesia, two main ways of pain control are used intra-operatively, one is opioids, the other is epidural. Many colleges prefer using epidural analgesia because it is potent and more effective , and also the benefits of stress block, less depression of breath. however, the epidural technique often causes more drop of blood pressure, especially in dehydrated patients. The investigators designed the trial to see if the benefit weigh out the potential risk of epidural in isolated hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

- adults aged 50-70 with isolated systolic hypertension .

Exclusion Criteria:

* age < 50 yr, ASA grade IV, severe cardiac or pulmonary insufficiency (FEV1 < 1 litre) , malignant hypertension, psychiatric illness (intake of psychiatric medication other than selective serotonin re-uptake inhibitors), diastolic blood pressure more than 110 mmHg. emergency surgery, coagulopathy, significant renal and hepatic dysfunction (creatinine > 50% or liver enzymes > 50% upper limit of normal values)

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Length of postoperative hospital stay | 5 weeks
cardiovascular morbidity | 2 weeks
respiratory morbidity | 2 weeks
postoperative renal failure | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dongxin Wang, MD, Study Chair — PKU 1st hospital
Locations (1):
- PKU 1st hospital, Beijing, Beijing Municipality, China